CLINICAL TRIAL: NCT00503009
Title: An Exploratory Study to Evaluate the Response of Salmeterol Plus Fluticasone vs Fluticasone Alone to Experimental Nasal Inoculation With Rhinovirus
Brief Title: Study Of RV-39 In Patients Who Also Have Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of data
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZA109895
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Rhinovirus; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: fluticasone propionate/salmeterol
- Arm 2 (Active Comparator)
  Interventions: Drug: fluticasone propionate
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol — comparator
  Other Names: fluticasone propionate
  Arms: Arm 1
Drug: fluticasone propionate — Comparator
  Arms: Arm 2
Drug: placebo — Placebo
  Arms: Arm 3

SUMMARY:
This study will last up to 9 weeks. Subjects will visit the clinic up to 14 times. Certain clinic visits will include a physical examination, lung function tests, inflammatory cell analysis from nasal secretions and/or sputum, and blood draws. Subjects will inhale an FDA approved virus through their nose which is known to cause the common cold. All study related medications and medical examinations will be provided at no cost to the subject. The drugs used in this study are approved for the age group under study.

ELIGIBILITY:
Inclusion Criteria:

* Have asthma for at least 3 months prior to the study.
* Have been using an allowed pre-study asthma therapy for at least 3 months prior to study.
* Demonstrate airway hyperresponsiveness following inhalation of bronchoconstrictor.
* Have a positive allergic status antibody test.

Exclusion Criteria:

* Have a history of life-threatening asthma.
* Been hospitalized for asthma within the 24 months prior to the study.
* Have certain conditions that would make study participation unsafe.
* The study doctor will evaluate other inclusion and exclusion criteria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZA109895 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects were randomized to one of two sputum induction groups (sputum induction, no sputum induction) and then stratified at a second randomization to one of three treatment groups (Fluticasone Propionate/Salmeterol [FSC 250/50] mcg twice a day [BID], Fluticasone Propionate [FP] 250 mcg BID, or Placebo BID).
Groups:
- FSC 250/50 mcg BID: Fluticasone Propionate/Salmeterol (FSC) (250/50 microgram) twice daily
- FP 250 mcg BID: Fluticasone Propionate (FP) (250 microgram) twice daily
- Placebo Diskus BID: Placebo twice daily
Period: Overall Study
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Started | 5 | 5 | 6
Completed | 4 | 3 | 3
Not Completed | 1 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID | Total
Number analyzed (Participants) | 5 | 5 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.4 (2.07) | 20.0 (1.00) | 23.0 (5.83) | 21.25 (3.8)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 5
  Male | 5 | 3 | 3 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5 | 2 | 4 | 11
  African American/African Heritage | 0 | 2 | 0 | 2
  American Indian/Alaskan Native/Native Hawaiian/Pac | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Cumulative Lower Respiratory Symptom Score Averaged Over Days 1-4
Description: The cumulative lower respiratory symptom score consisted of the summary of individual scores assessing cough, shortness of breath, chest discomfort, and wheezing based on the following scale: 0 (not present); 1=mild, clearly present; 2=moderately severe, uncomfortable; 3=severe (best possible score of 12; worst possible score of 0), interfering with sleep or activity. Due to the small sample size, efficacy measures were not analyzed.
Time Frame: Days 1 through 4
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Morning Peak Expiratory Flow (PEF) Averaged Over Days 1-4
Description: PEF measurements were collected via a study-issued electronic peak flow meter. Due to the small sample size, efficacy measures were not analyzed.
Time Frame: Days 1 through 4
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in the Morning Forced Expiratory Volume in One Second (FEV1) Averaged Over Days 1-4
Description: FEV1 measurements were collected via a study-issued spirometer. Due to the small sample size, efficacy measures were not analyzed.
Time Frame: Days 1 through 4
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Exhaled Nitric Oxide (eNO) Averaged Over Days 1-4
Description: eNO was measured using a study-issued monitor. Due to the small sample size, efficacy measures were not analyzed.
Time Frame: Days 1 through 4
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | FSC 250/50 mcg BID | FP 250 mcg BID | Placebo Diskus BID
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 250/50 mcg BID (N=5) | FP 250 mcg BID (N=5) | Placebo Diskus BID (N=6)
Heartburn (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the small sample size, efficacy measures were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.